CLINICAL TRIAL: NCT02240706
Title: A Phase I/II, Multicentre, Open-label, Dose Escalation and Randomized Trial of BI 836858 in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes
Brief Title: Phase I/II Trial to Investigate BI 836858 in Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1315.7; 2018-002177-21 (EudraCT Number)
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — BI 836858

ARMS (2):
- Arm B (Active Comparator): Best Supportive Care Alone
  Interventions: Procedure: Best Supportive Care
- Arm A (Experimental): BI 836858 plus Best Supportive Care
  Interventions: Procedure: Best Supportive Care; Drug: BI 836858

INTERVENTIONS:
Procedure: Best Supportive Care — At Discretion of the Investigator (Transfusions)
Drug: BI 836858 — Monotherapy with BI 836858
  Arms: Arm A

SUMMARY:
Phase I: To investigate maximum tolerated dose (MTD), safety and tolerability, pharmacokinetics, exploratory biomarker and efficacy of BI 836858 monotherapy in patients with low or intermediate-1 risk myelodysplastic syndromes (MDS) with symptomatic anemia. Phase II: To investigate safety and efficacy of BI 836858 plus Best Supportive Care compared to Best Supportive Care alone in low or intermediate-1 risk MDS patients with symptomatic anemia.

ELIGIBILITY:
Inclusion criteria:

* Documented diagnosis of Myelodysplastic Syndromes (MDS) according to World Health Organization (WHO) criteria that meets International Prognostic Scoring System (IPSS) classification of low or intermediate-1 risk disease at screening as determined by microscopic and standard cytogenetic analyses of the bone marrow and peripheral complete blood count (CBC).

  * Phase I dose escalation: patients who experienced Erythropoiesis-Stimulating Agents (ESA) treatment failure or do not qualify (serum erythropoietin level > 500 U) for ESA treatment, and are refractory to or not amenable or eligible for established MDS therapy (Hypomethylating Agents (HMA), lenalidomide)
  * Phase I expansion:

    * Expansion cohort 1 ("pre-treated"): patients who experienced ESA treatment failure or do not qualify (serum erythropoietin level > 500 U) for ESA treatment and are refractory to established MDS therapy (HMA and /or lenalidomide)
    * Expansion cohort 2 ("untreated"): patients who experienced ESA treatment failure or do not qualify (serum erythropoietin level > 500 U) for ESA treatment and who have not received prior HMA and/or lenalidomide (because not amenable or eligible for these treatments).
  * Phase II: patients who experienced ESA treatment failure or do not qualify (serum erythropoietin level > 500 U) for ESA treatment. For definition of further details of the phase II patients to be included the protocol will be amended based on Phase I results
* Patient is non-responsive to, refractory to, or intolerant of ESAs, or ESAs are contraindicated or unavailable, or a documented serum erythropoietin level of > 500 U/L.
* Eastern Cooperative Oncology Group (ECOG) Performance Status <=2.
* Age >= 18 years.
* Written informed consent which is consistent with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines and local legislation.

Exclusion criteria:

* Patient with IPSS category of Int-2 or high-risk MDS.
* Phase II only: Patients with a deletion 5q cytogenetic abnormality.
* Treatment within 28 days prior to Cycle 1 Day 1 with: i) long acting erythropoiesis stimulating agents, ii) long acting Granulocyte colony-stimulating factor (G-CSF), iii) granulocyte- macrophage colony stimulating factor (GM-CSF), iv) 5-aza, lenalidomide or decitabine, or v) iron chelation and within 14 days prior to Cycle 1 Day 1 with short acting erythropoiesis stimulating agents and short acting G-CSF.
* Patient previously received allogeneic bone marrow or stem cell transplantation.
* Second malignancy currently requiring active therapy (except for hormonal/antihormonal treatment, e.g. in prostate or breast cancer).
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) > 2.5 times the upper limit of normal (ULN).
* Bilirubin >1.5 mg/dL, except for Gilbert's Syndrome or hemolysis.
* Serum creatinine >2.0 mg/dL.
* Known human immunodeficiency virus (HIV) infection and/or active hepatitis B infection (defined as presence of Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA).
* Presence of concomitant intercurrent illness, or any condition which in the opinion of the Investigator, would compromise safe participation in the study, e.g. active severe infection, unstable angina pectoris, new onset of exacerbation of a cardiac arrhythmia.
* Psychiatric illness or social situation which in the opinion of the Investigator would limit compliance with trial requirements.
* Patient receiving concomitant therapy, which in the opinion of the Investigator is considered relevant for the evaluation of the efficacy or safety of the trial drug.
* Female patients of childbearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial and for 6 months after the last administration of BI 836858, i.e. combination of two forms of effective contraception (defined as hormonal contraception, intrauterine device, transdermal patch, implantable or injectable contraceptive, bilateral tubal ligation etc.).

Women of childbearing potential are defined as females who:

* Have experienced menarche and
* Are not postmenopausal (12 months with no menses without an alternative medical cause) and
* Are not permanently sterilized (e.g. hysterectomy, bilateral oophorectomy or bilateral salpingectomy

  * Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second effective method of contraception (defined as hormonal contraception, intrauterine device, condom with spermicide, etc.) during the trial and for 6 months after the last administration of BI 836858.
  * Pregnant or nursing female patients.
  * Treatment with another investigational agent under the following conditions:
* Within two weeks (4 weeks for biologics) of first administration of BI 836858, or if the half-life of the previous product is known, within 5 times the half-life, whichever is longer.
* Patient has persistent toxicities from prior MDS therapies which are determined to be relevant by the Investigator.
* Concomitant treatment with another investigational agent while participating this trial.

  * Chronic use, as defined by > 2 weeks of a corticosteroid agent that is >= 20 mg/day of prednisone or its equivalent, within 4 weeks prior to first administration of BI 836858.
  * Treatment with an immunomodulatory agent within 4 weeks prior to first administration of BI 836858.
  * Patient received prior treatment with a CD33 antibody.
  * In the opinion of the Investigator patient is unable or unwilling to comply with the protocol.
  * Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- United States (3):
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cleveland Clinic, Cleveland, Ohio
- Germany (2):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a phase I/II, multicenter, open-label, dose escalation and randomized trial of BI 836858 in patients with low or intermediate-1 risk myelodysplastic syndromes.
Pre-assignment Details: Subjects were screened for eligibility prior to participation. They attended a specialist site which ensured that they strictly met all eligibility criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 836858 20 mg (Phase I): All patients were administered doses of BI 836858, 20 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 40 mg (Phase I): All patients were administered doses of BI 836858, 40 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 80 mg (Phase I): All patients were administered doses of BI 836858, 80 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 160 mg (Phase I): All patients were administered doses of BI 836858, 160 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 320 mg (Phase I): All patients were administered doses of BI 836858, 320 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 + Best Supportive Care (BSC) (Phase II): All patients were planned to be administered doses of BI 836858, recommended phase 2 dose (RP2D) together with best supportive care (BSC) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- Best Supportive Care (BSC) Only (Phase II): All patients were planned to be administered best supportive care (BSC) including red blood cell transfusion, platelet transfusion and iron chelation therapy.
Period: Overall Study
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I) | BI 836858 + Best Supportive Care (BSC) (Phase II) | Best Supportive Care (BSC) Only (Phase II)
Started | 3 | 3 | 6 | 4 | 11 | 0 (No patients were enrolled in the Phase II part due to strategic reasons.) | 0 (No patients were enrolled in the Phase II part due to strategic reasons.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 4 | 11 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 2 | 2 | 5 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Refused to continue taking medication | 0 | 1 | 3 | 1 | 2 | 0 | 0
Not completed — Insurance billing concerns | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (5.57) | 75.0 (6.24) | 73.8 (16.41) | 68.3 (12.18) | 75.6 (5.08) | 73.6 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 2 | 4 | 7
  Male | 3 | 3 | 5 | 2 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 4 | 11 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 4 | 11 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: The MTD is defined as the highest dose of BI 836858 with less than 25% risk of the true dose-limiting toxicity (DLT) rate being above 33% during the MTD evaluation period. MTD determination will be based on a Bayesian logistic regression model with overdose control.
  For any dose-escalation cohort, at least 3 patients (pts) will be required. However, in the case that only 2 pts are evaluable and neither has experienced a DLT within the first cycle (2 administrations - 28 days), then dose-escalation can occur based on these 2 pts. After all pts in a cohort have either experienced a DLT or have been observed for at least one cycle (2 administrations - 28 days) without experiencing a DLT, the Bayesian model will be updated with the newly accumulated data.
  The MTD may be considered reached if either the posterior probability of the true DLT rate in the target interval (16%-33%) is above 50%, or at least 12 pts have been treated at MTD, including the two expansion cohorts.
Time Frame: From the first administration of BI 836858 to start of the third administration of BI 836858, excluding the day of the third administration of BI 836858, up to 28 days
Population: As the study was prematurely discontinued, recruitment of participants into the dose escalation part was not fully completed. No formal MTD was determined.
Groups:
- BI 836858: Treatment group "BI 836858" comprises all dose cohorts during the dose escalation phase, that is, "BI 836858 20 mg", "BI 836858 40 mg", "BI 836858 80 mg", "BI 836858 160 mg" and "BI 836858 320 mg".
  All patients were administered doses of BI 836858, by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
Arm/Group | BI 836858
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) (Phase I)
Description: Dose Limiting Toxicity (DLT):
  * Grade (G) ≥ 3 (CTCAE 4.0), non disease-related, non-hematologic adverse events (AE), except:
    * Laboratory abnormality, not significant by investigator or resolves spontaneously or can be recovered with appropriate treatment (T) within 5 d
    * Neutrophils (NP) <500 /microliters (μL) at T start, febrile neutropenia with NP <500 /μL or infection with NP <500 /μL will not constitute a DLT if they can be recovered with appropriate T within 14 d
  * Inability to deliver study drug full dose according to the assigned dose level within cycle 1 due to drug-related AEs
  * Absence of hematological recovery as following:
    * NPs: G 4 (if G 0/1 at baseline (BL)) OR <100 /μL and decrease of >75% from BL (if G ≥2 at BL) for >7 d
    * Platelets: G 4 (if G 0/1 at BL) OR < 10000/μL for >7 d and decrease of >75% from BL (if G ≥2 at BL)
  * T delay of ≥4 weeks of start of Cycle 2 --If Cycle 2 is not started until 57th d as a result of drug related AE, it is considered as DLT
Time Frame: as for outcome 1
Population: MTD evaluation set: All patients who were documented to have initiated at least one dose of BI 836858 and who have not been replaced for the MTD evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 2 | 3 | 6 | 4 | 9
Participants | 0 | 0 | 1 | 0 | 2

3. Secondary Outcome: Number of Patients With Red Blood Cell (RBC) Transfusion Independency (Phase I)
Description: Number of patients with red blood cell (RBC) Transfusion Independency is presented.
  Red blood cell (RBC) transfusion independence and platelet transfusion independence will be evaluated in patients who are transfusion dependent at baseline. Percentages will be calculated using all treated patients as the denominator.
  A patient is considered transfusion independent at baseline if the patient has had no transfusions during the 56 days prior to and including the first day of treatment. Otherwise, the patient is considered to be transfusion dependent.
  A patient is considered transfusion independent if the patient has had no transfusions over the course of ≥ 56 consecutive days.
Time Frame: From first administration of BI 836858 until discontinuation of the treatment. Up to 168 days (6 cycles, each of 28 days)
Population: Treated set (TS): The TS included all patients who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Patients With Hematologic Improvement Neutrophils (HI-N) (Phase I)
Description: Number of patients with hematologic improvement neutrophils (HI-N) is presented.
  The HI will be evaluated in patients with abnormal pretreatment values defined as follows:
  Neutrophil response (HI-N) - Patients with a pretreatment neutrophil count <1 x 10^9/liters (L) demonstrate a neutrophil response if they have an at least 100 percent increase and an absolute increase >0.5 x 10^9/L.
Time Frame: From first administration of BI 836858 until HI-N, up to 168 days (6 cycles, each of 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Hematologic Improvement Platelets (HI-P) (Phase I)
Description: Number of patients with hematologic improvement platelets (HI-P) is presented.
  The HI will be evaluated in patients with abnormal pretreatment values defined as follows:
  Platelet response (HI-P) - Patients with a pretreatment platelet count <100 x 109/Liters (L) demonstrate a platelet response if there is an absolute platelet increase of ≥30 x 109/L for patients starting with >20 x 109/L platelets. For those with an increase from 10 x 109/L to >20 x 109/L must have an increase of at least 100 percent.
Time Frame: From first administration of BI 836858 until HI-P, up to 168 days (6 cycles, each of 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Hematologic Improvement Erythroid (HI-E) (Phase I)
Description: Number of patients with hematologic improvement erythroid (HI-E) is presented.
  The HI will be evaluated in patients with abnormal pretreatment values defined as follows:
  Erythroid response (HI-E): Patients with a pretreatment hemoglobin <11 grams per deciliters (g/dL) demonstrate erythroid response if their hemoglobin increases by ≥1.5 g/dL for at least eight weeks, and there is a reduction in the units of red cell transfusions by an absolute number of at least four red cell transfusions per eight weeks compared with the pretreatment transfusion number in the previous eight weeks. Only red cell transfusions given for a hemoglobin ≤9 g/dL pretreatment will count in the red cell transfusion response evaluation.
Time Frame: From first administration of BI 836858 until HI-E, up to 168 days (6 cycles, each of 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Time to HI-E Response (Phase I)
Description: Time to HI-E response is defined only for patients who achieve a HI-E response as follows: Time to HI-E response [days] = date of first assessment indicating HI-E response - date of first administration of trial medication + 1.
Time Frame: From first administration of BI 836858 until HI-E response, up to 168 days (6 cycles, each of 28 days)
Population: Treated set (TS): The TS included all patients who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses. Only patients who showed a HI-E response were included.
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Patients With Mean Hemoglobin Increase ≥ 1.5 g/dL (Phase I)
Description: Number of patients with mean hemoglobin increase ≥ 1.5 grams per deciliters (g/dL) is presented.
  Mean hemoglobin increase ≥ 1.5 g/dL - Proportion of subjects achieving hemoglobin (Hgb) increase from baseline ≥ 1.5 g/dL over any consecutive 56-day period in absence of Red blood cell (RBC) transfusions.
Time Frame: Up to 48 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11
Participants | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Duration of Response (RBC Transfusion Independency, HI-N, HI-P, HI-E or Objective Response) (Phase I)
Description: Defined only for patients who achieve complete Response (CR) or marrow complete response (mCR) or RBC Transfusion independency (TI), measured from first date of achieving response until date of relapse. Date of relapse will be earliest of dates of disease assessment (blood sample, bone marrow sample, or clinical assessment) in which relapse was observed. For patients who die or are lost to follow-up without documented relapse, response duration will be censored, respectively, on date of death, regardless of cause, or on date of last disease assessment for patients who are alive when lost to follow-up. Duration of Response [days] = date of outcome - date of first assessment indicating CR or mCR or RBC TI after first administration of trial medication + 1.
Time Frame: From the first date of achieving a response until the date of relapse, up to 168 days (6 cycles, each of 28 days)
Population: Treated set (TS): The TS included all patients who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses. Only patients who had achieved complete response (CR) or marrow complete response (mCR) or RBC Transfusion independency (TI) were included.
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Patients With Overall Objective Response (OR) [Complete Response (CR), Partial Response (PR), and Hematologic Improvement (HI)] (Phase I)
Description: Number of patients with overall Objective Response (OR) [Complete Response (CR), Partial Response (PR), and Hematologic Improvement (HI)] is presented.
  Overall Objective Response is defined as Complete Response (CR), Partial Response (PR), HI-N, HI-P, or HI-E. A patient's " Overall Objective Response " = "Yes" if one of these responses was reported at least once throughout the trial.
  CR defined as: -Bone marrow: <5 % blasts with normal maturation of all cell lines (Dysplastic changes should consider the normal range of dysplastic changes), persistent dysplasia will be noted; -Peripheral blood: Hgb > 11 grams per deciliters (g/dL), Platelets >100 x 109/liters (L), Neutrophils > 1.0 x 109/L, Blasts 0 % PR defined as: -All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by >50 % to pre-treatment but still >5 %, Cellularity and morphology not relevant.
  HI Definition see other endpoints.
Time Frame: From first administration of BI 836858 until overall objective response, up to 168 days (6 cycles, each of 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836858 20 mg (Phase I) | BI 836858 40 mg (Phase I) | BI 836858 80 mg (Phase I) | BI 836858 160 mg (Phase I) | BI 836858 320 mg (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 11
Participants | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Patients With Red Blood Cell (RBC) Transfusion Independency (Phase II)
Description: Red blood cell (RBC) transfusion independence and platelet transfusion independence will be evaluated in patients who are transfusion dependent at baseline. Percentages will be calculated using all treated patients as the denominator.
  A patient is considered transfusion independent at baseline if the patient has had no transfusions during the 56 days prior to and including the first day of treatment. Otherwise, the patient is considered to be transfusion dependent.
  A patient is considered transfusion independent if the patient has had no transfusions over the course of ≥ 56 consecutive days.
Time Frame: as for outcome 3
Population: No patients were enrolled in the Phase II part. The company decided to stop the clinical development of BI 836858 prematurely during the Phase I expansion cohort stage for strategic reasons.
Arm/Group | BI 836858 + Best Supportive Care (BSC) (Phase II) | Best Supportive Care (BSC) Only (Phase II)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first administration of BI 836858 until end of residual effect period (REP), up to 198 days. For all-cause mortality from first administration of BI 836858 until end of follow-up, up to 198 days + 6 months follow-up.
Description: Treated set (TS): The TS included all subjects who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Groups:
- BI 836858 20mg: All patients were administered doses of BI 836858, 20 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 40mg: All patients were administered doses of BI 836858, 40 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 80mg: All patients were administered doses of BI 836858, 80 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 160mg: All patients were administered doses of BI 836858, 160 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
- BI 836858 320mg: All patients were administered doses of BI 836858, 320 milligrams (mg) by a rate-controlled intravenous infusion on day 1 and on day 15 of a 28-day cycle for a duration of 4 cycles. All infusions were to be started at a rate of 10 mL/h. The infusion rate was to be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient.
Arm/Group | BI 836858 20mg | BI 836858 40mg | BI 836858 80mg | BI 836858 160mg | BI 836858 320mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 1/6 | 0/4 | 3/11
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 3/6 | 0/4 | 6/11
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 4/4 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836858 20mg (N=3) | BI 836858 40mg (N=3) | BI 836858 80mg (N=6) | BI 836858 160mg (N=4) | BI 836858 320mg (N=11)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836858 20mg (N=3) | BI 836858 40mg (N=3) | BI 836858 80mg (N=6) | BI 836858 160mg (N=4) | BI 836858 320mg (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 3
Monocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2 | 1 | 1
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 5 | 4 | 7
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Carotid bruit (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 2 | 1 | 3
Platelet count decreased (Investigations) | 0 | 1 | 1 | 1 | 1
QRS axis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Development of BI 836858 was discontinued (strategic decision) during the Phase I Expansion cohort stage. No patients were enrolled in the Phase II part.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT02240706/SAP_000.pdf
  • Study Protocol (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT02240706/Prot_001.pdf